CLINICAL TRIAL: NCT01598558
Title: Assessing Response to Treatment in Non-Hodgkin's Lymphoma Patients Using 64Cu-DOTA-Rituximab PET/CT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual issues - Low Accrual
Sponsor: Sanjiv Sam Gambhir (Other)
Responsible Party: Sponsor-Investigator, Sanjiv Sam Gambhir, Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LYMIMG0002; 8556 (Other: Stanford IRB)
Record Dates: First submitted 2012-02-10; First posted 2012-05-15 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 64Cu-DOTA (Experimental): Subjects will be injected with less than 14 mCi of 64Cu-DOTA-Rituximab. This is a slow infusion, done over 20 minutes.
  Interventions: Drug: Cu-64 Rituximab

INTERVENTIONS:
Drug: Cu-64 Rituximab — Up to 14 mCi, iv
  Other Names: Genentech/MIPS

SUMMARY:
Rituximab is an antibody targeted against the CD20 antigen found primarily on B-cells. Therefore, an imaging agent targeting CD20 expression may provide a more accurate evaluation of extent of disease and response to therapy than the current standard of care, F-18 FDG PET/CT.

The main purpose of the study is to investigate a new PET/CT imaging probe for detection and follow up of lymphoma. Following are the 3 aims of the study: a) Phase I testing in lymphoma patients of Cu-64 labelled Rituxan for defining normal tracer biodistribution, stability, pharmacokinetics and radiation dosimetry; b) comparison of Cu-64 Rituxan and F-18 FDG PET/CT in lymphoma patients; c) evaluation of changes in uptake of Cu-64 Rituxan in response to rituximab-based treatment in CD20-positive B-cell NHL

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of CD20-positive B-cell NHL and a staging 18F FDG PET/CT prior to the 64Cu-DOTA-Rituximab PET/CT
* Patients must understand and voluntarily sign an Informed Consent form after the contents have been fully explained to them
* Patients must be scheduled for rituximab-based therapy
* Patients must be older than 18-year-old

Exclusion Criteria:

* Patients who cannot complete a PET/CT scan
* Pregnant women
* Patients participating in other research protocols will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in pre and post treatment SUV max value on the 64CU-DOTA-Rituximab PET/CT and 18F FDG PET/CT | baseline and 6 weeks
  Pre- and post-treatment tumor SUVmax value on the 64Cu-DOTA-Rituximab PET/CT and 18F FDG PET/CT, and resulting EORTC-based classification of patients as responding or not responding to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Gambhir, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States